CLINICAL TRIAL: NCT04858620
Title: A Randomized Placebo Control Trial to Evaluate the Efficacy of Xlear vs. Placebo for Acute COVID-19 Infection
Brief Title: A Study to Evaluate the Efficacy of Xlear vs. Placebo for Acute COVID-19 Infection
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Period Ended / Not Completed
Sponsor: Larkin Community Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LCH-3-032020
Record Dates: First submitted 2021-02-04; First posted 2021-04-26 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Masking to care providers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- No treatment (No Intervention)
- Treatment (Experimental)
  Interventions: Drug: Xlear Nasal Spray
- Placebo (Placebo Comparator): Saline nasal spray, 2 puffs per nostrils, every 6 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xlear Nasal Spray — Xylitol plus Grapefruit Seed Extract (Xlear) nasal spray, 2 puffs per nostrils, every 6 hours
  Arms: Treatment
Drug: Placebo — Saline nasal spray, 2 puffs per nostrils, every 6 hours
  Arms: Placebo

SUMMARY:
This study aims to find out the efficacy of Xlear nasal spray as an adjunct medication against COVID-19. This encompasses reduction in the number of days to negativization via nasal swab PCR from the average 14 days and early improvement of symptoms.

DETAILED DESCRIPTION:
Patients will be informed about the study including potential risk and benefits. Once written informed consent are obtained, patients will undergo a brief screening period to determine eligibility for the study. Once eligibility is confirmed, eligible patients will be placed in a randomized placebo control manner. Patient will be assigned to Xlear (2 puffs per nostrils, every 3-4 hours a day) or placebo. Patient will be followed for 1 week. Inflammatory markers will be obtained on Day 4 and repeat COVID-19 Reverse Transcriptase PCR (RT PCR) on Day 7. Follow up will be done on Day 14 for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of ages 18 to 90 years of both sexes
2. With positive SARS-CoV-2 carriage confirmed by nasopharyngeal PCR
3. Signed informed consent
4. Mild symptoms: Minimum respiratory symptoms or asymptomatic plus positive test
5. Moderate symptoms: Respiratory symptoms such as cough, mild shortness of breath with mild oxygen desaturation(room air SpO2 <92% and >88% or <88% corrected to >92% with 2 liters of oxygen)

Exclusion Criteria:

1. Patient with very low viral load (threshold cycle [Ct] > 25 per PCR).
2. Known hypersensitivity to one of the constituents, particularly to xylitol or grapefruit seed extract (GSE)
3. Under 18 years of age
4. Women of childbearing age who are pregnant, breastfeeding mothers, and intend to become pregnant during the study period; unwilling/unable to take a pregnancy test.
5. Unable to provide informed consent or decline to consent or unwillingness to adhere to the Standard of Care protocol.
6. Patients with severe symptoms -Hypoxia (SpO2 <88% not corrected by 2 liter non-concentrated oxygen) plus severe shortness of breath
7. History of immunodeficiency or are currently receiving immunosuppressive therapy
8. Have had a planned surgical procedure within the past 12 weeks.
9. Already part of this trial, recruited at a different hospital.
10. Patient unable to perform oro-nasopharyngeal decolonization
11. Patients with acute exacerbation of severe comorbidities like heart disorders Chronic Obstructive Pulmonary Disease (COPD), Heart Failure New York Heart Association (NYHA) Class 3 and 4 and/or diseases with severe oxygenation problems
12. Patients on Remdesivir and/or other clinical trials.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Hasten baseline reactive to non-reactive on COVID 19 RT PCR | Baseline and 7 days
  The COVID 19 RT PCR is the gold standard in the detection of COVID 19 in patients. With the average time to negativization being 14 days. This study aims to reduce the reactivity to 7 days.

SECONDARY OUTCOMES:
Change of symptoms | Baseline and 7 days
  Monitor changes in daily symptoms for COVID 19 positive patients using Symptom Assessment Scale (SAS). Symptoms are classified as Mild, Moderate, Severe.
Change of symptoms | Baseline and 7 days
  Monitor changes in daily symptoms for COVID 19 positive patients using Visual Analogue Scale (VAS). Symptoms are classified using a a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Change of symptoms | Baseline and 7 days
  Monitor changes in daily symptoms for COVID 19 positive patients using Numerical Rating Scale (NRS). Symptoms are classified from 1-10, with 1 being no symptoms and 10 worst symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Larkin Community Hospital, Miami, Florida, United States